CLINICAL TRIAL: NCT05939830
Title: Omission of Axillary Lymph Node Dissection in Breast Cancer Patients With Axillary Pathological Complete Response After Neoadjuvant Systemic Therapy
Brief Title: Omission of ALND in Breast Cancer Patients With Axillary pCR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jue Wang, Prof., The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SrLNB
Record Dates: First submitted 2023-07-01; First posted 2023-07-11 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Axillary Lymph Node Dissection; Pathological Complete Response; Neoadjuvant Systemic Therapy; Breast Cancer; Axillary Lymph
Keywords: Breast Cancer; Neoadjuvant Systemic Therapy; Axillary Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Omit ALND (Experimental): Omitting Axillary Lymph Node Dissection (ALND) in SrLNB-proven axillary complete response patients.
  Finishing regional lymph node irradiation (RNI) including the axilla after surgery.
  Interventions: Procedure: Stained region Lymph Node Biopsy (SrLNB); Radiation: Regional lymph node radiotherapy (RNI) including the axilla

INTERVENTIONS:
Procedure: Stained region Lymph Node Biopsy (SrLNB) — Before NST, carbon nanoparticles suspension would be injected into the cortex of positive lymph nodes for staining under ultrasound guidance. Marked lymph nodes will be removed and biopsied after NST.
Radiation: Regional lymph node radiotherapy (RNI) including the axilla — RNI including the axilla covers the supraclavicular region and entire axillary lymphatic drainage area (region I, II and III) ,and is at a dose of 50 Gy/25 times, with additional prophylactic irradiation of the internal breast lymphatic drainage area for eligible patients.

SUMMARY:
This prospective, single-arm, phase II trial studies axillary lymph node dissection (ALND) to see if it can be safely omitted in breast cancer patients with axillary pathological complete response (pCR) after neoadjuvant systemic therapy (NST). Breast cancer patients with biopsy-proven positive axillary lymph nodes at initial diagnosis, and converted to negative after NST, which is confirmed by Stained region Lymph Node Biopsy(SrLNB), will be enrolled in the study. In other words, a total of 92 patients will be exempted from ALND after SrLNB, and afterwards complete regional node irradiation (RNI) including the axilla. They will also undergo adjuvant chemotherapy, targeted therapy, endocrinotherapy after surgery. These patients will be followed up in the next three years for local-regional recurrence and long-time survival outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged between 18 and 70 years;
2. Pathologically confirmed invasive breast cancer (regardless of pathological type) with a clinical stage cT1-3;
3. Pathologically confirmed positive axillary lymph nodes with a clinical stage of N1-3;
4. Receiving a full course of neoadjuvant therapy (including neoadjuvant chemotherapy, neoadjuvant targeted therapy, neoadjuvant immunotherapy);
5. Positive axillary lymph nodes successfully stained by carbon nanoparticles injection;
6. All patients are required to undergo immunohistochemical staining for Estrogen Receptor (ER), Progesterone Receptor (PR), human epidermal growth factor receptor 2 (HER2), Ki- 67 proliferation index, and further fluorescence in situ hybridization (FISH) should be performed in HER2 2+ cases;
7. Preoperative clinical assessment (including physical examination, imaging, with or without nomogram assessment) suggests positive axillary lymph nodes converted to negative (ycN0);
8. ECOG score 0 - 1;
9. Patients voluntarily participated in this study and signed the informed consent form

Exclusion Criteria:

1. Bilateral breast cancer;
2. Breast cancer during lactation period or pregnancy;
3. Physical examination or imaging examination confirmed presence of distant metastases;
4. Previous history of malignant tumor;
5. History of previous surgery on the affected axilla; or history of surgery affecting the function of the upper extremity;
6. History of radiation therapy to the breast or chest;
7. Positive incision margins for breast-conserving surgery/mastectomy;
8. Positive results of intraoperative rapid freeze pathology (including isolated tumor cells and micrometastases) for SrLNB (ypN+);
9. Those who unable to complete the full course of follow-up adjuvant therapy as prescribed for various reasons;
10. Aspartate transaminase (AST) and alanine transaminase (ALT) ≥ 1.5 times the upper limit of normal, alkaline phosphatase（ALP） ≥ 2.5 times the upper limit of normal, total bile ≥ 1.5 times the upper limit of normal, serum creatinine ≥ 1.5 times the upper limit of normal; Left Ventricular Ejection Fractions (LVEF) < 50% in cardiac ultrasound;
11. Severe coagulation dysfunction, serious systemic disease, or uncontrolled infection;
12. Without personal freedom and independent civil capacity;
13. Those with mental disorders, addictions, who were not eligible for enrollment in the judgment of the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
iDFS: invasive Disease-Free Survival after breast surgery | Up to 3 years after surgery
  Time interval from the surgery to invasive local-regional recurrence, distant metastasis, contralateral invasive breast cancer, or death from any cause.

SECONDARY OUTCOMES:
LRR: Local-Regional Recurrence after breast surgery | Up to 3 years after surgery
  This includes both local and regional recurrences. Local recurrence is defined as recurrence in the ipsilateral breast, chest wall, skin or surgical scar. Regional recurrence is defined as recurrence in the affected lymphatic drainage area, including the axilla, supraclavicular region, subclavicular region, and internal mammary node area.
BCRL: Breast Cancer Related Lymphedema | Up to 3 years after surgery
  Objective evaluation of upper limb lymphedema by arm circumference and bioelectrical impedance measurement. In our study, BCRL is diagnosed in two ways：① Relative Volume Change (RVC ) >10% in the affected upper extremity. ②Bioelectrical impedance technology: the impedance ratio is defined as the ratio of the impedance of the healthy upper limb to the impedance of the affected upper limb, and BCRL is diagnosed when the patient's impedance ratio is higher than the mean + 2 standard deviations (SD) of healthy controls. When the two measurements are inconsistent, the former results shall prevail.
Quality of life (QoL) | Up to 3 years after surgery
  Patients' subjective assessment of quality of life (QoL) using the Functional Assessment of Cancer Therapy-Breast (FACT-B) . FACT-B is divided into 36 items in 5 domains, namely: physical status (7 items), social/family status (7 items), emotional status (6 items), functional status (7 items) and additional concerns, and each item is classified into five levels: not at all (0), somewhat (1), somewhat (2), fairly (3) and very much (4). Positive items were scored directly from 0 to 4, while negative items (i.e., the larger the number of response options, the worse the quality of life) were scored in reverse. The total score of FACT-B scale ranges from 0 to 144, a higher score means a better quality of life for the patient.
Patient-reported arm morbidity | Up to 3 years after surgery
  Patients' subjective assessment of lymphedema using the Quick Disability of the Arm, Shoulder, and Hand (Quick DASH) questionnaires，Quick DASH consists of 11 items, and is a self-rating scale of daily functioning including social functioning and physical activity and upper extremity symptoms. Each item is divided into 5 levels, and the patient's score is calculated as score = [(patient score/number of response items) - 1] × 25, with a total score of 0 to 100, and the higher the score, the greater the degree of upper limb dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma L, Chen R, Wang M, Li X, Zheng R, Wang L, Ding J, Yao H, Gong Y, Wang Y, Sheng X, Wang J, Zha X. Omission of axillary lymph node dissection in patients with breast cancer with axillary pathological complete response confirmed by stained region lymph node biopsy after neoadjuvant systemic therapy (SrLNB study): study protocol for a single-arm, single-centre, phase-II trial. BMJ Open. 2025 Mar 31;15(3):e092563. doi: 10.1136/bmjopen-2024-092563. PMID 40164484